CLINICAL TRIAL: NCT04652622
Title: Use of a Novel Digital Therapeutic Intervention for the Management of Delirium in the Acute Care Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Collaborators: BC Support Unit (Other); Royal Columbian Hospital Foundation (Other); Mitacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FHREB 2020-091
Record Dates: First submitted 2020-11-17; First posted 2020-12-03 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Delirium
Keywords: digital therapeutic; behavioral; critical care; behavior modification
MeSH Terms: conditions — Delirium; Behavior

STUDY DESIGN:
Intervention Model Description: participants will be randomized to either exposure to the intervention arm in conjunction with standard care or the control arm and will receive standard care alone
Who Masked: Outcomes Assessor
Masking Description: data will be blinded for analysis but the study is open label due to the nature of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants will receive 4 hours of exposure to the Mindful Garden digital therapeutic platform in addition to standard care
  Interventions: Device: Mindful Garden
- Control Arm (No Intervention): Participants will be monitored over a 4 hour period of standard care interventions

INTERVENTIONS:
Device: Mindful Garden — Mindful Garden is an interactive digital behavior modification platform utilizing inbuilt sensors and screen based delivery system. The platform delivers calming visual output of real nature video layered with hyper-real animations of growing and receding flowers and butterflies in flight in a volume directly responsive to measured patient activity. Patient movement and vocalization are the surrogate markers for agitation and using proprietary algorithms drive onscreen content.
  Arms: Intervention arm

SUMMARY:
Delirium is a condition of fluctuating confusion and agitation that affects as many as 80% of patients in critical care. Hyperactive delirium consumes a significant amount of clinical attention and resources due to the associated psychomotor agitation. Patients can become aggressive or combative putting both themselves and healthcare workers at risk of harm. Delirium has been linked to an increased risk of death and poor overall outcomes. Management largely relies on the use of potentially toxic medications and physical restraints despite limited proof of success of these interventions. Our research group will study the use of a novel interactive digital therapeutic behavior modification platform aimed at reducing anxiety and agitation associated with hyperactive delirium. We hypothesize that Use of the Mindful Garden behavioral modification platform will result in normalization of agitation and delirium scores when used for the management of delirium associated agitation in the adult delirious acute care population compared to standard care alone.

DETAILED DESCRIPTION:
Mindful Garden is a digital behavior modification platform that utilizes screen based delivery systems and sensor technologies. Mindful Garden delivers real 2-dimensional nature video layered with hyper-real 3-dimensional animations of growing and receding flowers and butterflies in flight which aims to reduce anxiety and agitation in the delirious critical care population. In doing so, normalization of agitation and delirium scores may be achieved as well as a reduction in reliance on pharmacological interventions and the use of physical restraints, which have been linked to adverse outcomes and significant side effects.

Participants with a diagnosis of hyperactive delirium in acute care inpatient units will be randomized to receive 4 hours of exposure to the MG platform in addition to standard care or to the control arm of monitoring with standard care only for the same time period.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age >18yrs)
* Admitted to the Royal Columbian Hospital
* RASS +1 or greater for 2 assessments 1 hour apart within the 24-hour period directly prior to study enrollment and persisting at the time of enrollment
* Demonstrated incidence of at least 2 PRN medication events for the management of delirium-associated agitation in the preceding 24 hours and/or infusion of psycho- active medication for the management of delirium (eg: dexmeditomodine)
* ICDSC greater than or equal to 4 at time of enrollment or CAM positive

Exclusion Criteria:

* Planned procedure or test that precludes participation in the full 4-hour study session
* Unable to see (visual impairment such as documented blindness, ongoing inability to keep eyes open or documented or assessed inability to focus, track or maintain visual contact for extended periods as determined by recruitment personnel)
* Significant uncontrolled pain with a Verbal Pain scale of 5/10 or greater or a Clinical Pain Observation Tool >4 despite intervention at the time of enrollment.
* RASS of 0 to -5 at study enrollment indicating patient is awake and calm or sedated
* Refusal for participation by the participant's responsible physician or request to not retain data by participants substitute decision maker
* Currently enrolled in any other research study involving drugs or devices which could impact on the outcomes of interest, as evaluated by the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Agitation scores | 5 hours
  Richmond Agitation Sedation Score is a validated and standardized scoring system ranging from -5 (deeply sedated) to 0 (awake and calm) to +4 (combative). Scores are measured hourly from study start, one hour post intervention and at the start of the following nursing shift.

SECONDARY OUTCOMES:
Use of unscheduled medications for the management of delirium associated agitation | 4 hours
  Incidence of unscheduled or "PRN" medication use for the management of delirium associated agitation throughout the 4 hour study period
Delirium Scores | 4 hours
  Delirium scores will be measured using the Intensive Care Delirium Screening Checklist. Delirium score is a range of zero to 8 with scores above or equal to 4 being diagnostic for the presence of delirium and higher scores being indicative of added severity of symptoms. Intensive Care Delirium Screening Checklist will be measured at study initiation, after 2 hours, at study completion (4 hours) and the start of the following nursing shift
Richmond Agitation Sedation Scale of zero | 4 hours
  Proportion of patients achieving a Richmond Agitation Sedation Scale score of zero throughout the study period. Score range is -5 to +4 with a score of zero indicating the patient is awake and calm. Negative scores indicate deeper sedation, positive scores reflect agitation
Physical Restraint Use | 4 hours
  Proportion of participants with physical restraints in use throughout the study period and the length of time of restraints in use
Incidence of Unplanned Line removal | 4 hours
  Incidence of unplanned removal of lines or tubes by the study participant (endotracheal tubes, nasogastric tubes, oral-gastric tubes, central venous lines, peripheral intravenous lines, urinary catheters, arterial lines) throughout the study period.
PRN medication use in the 2 hours post study | 2 hours
  Incidence of unscheduled medication administration for the management of delirium behaviors in the 2 hours following the study or intervention period.
Movement Count Average | 4 Hours
  Those in the intervention arm will have generated activity logs stored within the device units. The movement count average is calculated by comparing the difference in pixel density from the previous frame to the current one. The resulting value is then averaged over the collected frames and returned as a decimal percentage of change. Values are between 0 and 1 with 0 showing the lowest amount of activity and one the highest
Physiological data | 4 hours
  Basic physiological data will be collected and analyzed from nursing records and for a smaller proportion directly from telemetry monitors where available to compare between arms as well as to evaluate trends over the course of the study period. Parameters include heart rate, mean arterial blood pressure, respiratory rate, oxygen saturation and use of vasopressors
heart rate variability | 6 hours
  For a small subset of the overall population ECG data will be collected to assess differences in heart rate variability between study arms measured as pNN50 and RMMSD. Five minute ECG recordings will be taken hourly starting one hour before the study period until one hour post timed to match agitation and delirium scores

OTHER OUTCOMES:
Survey of caregivers | 4 hours
  a 5 question survey of caregivers will be conducted using a 9 point Likert scale evaluating the ease of use of the intervention and acceptability of the intervention. On the scale 1 indicates strongly disagree to 9 indicating strongly agree, 5 being neutral. The questionnaire will be conducted at the end of the study period where possible
Survey of family members | 4 hours
  a 5 question survey of family members if present during exposure to the intervention will be conducted using a 9 point Likert scale evaluating acceptability of the intervention. On the scale 1 indicates strongly disagree to 9 indicating strongly agree, 5 being neutral

CONTACTS AND LOCATIONS:
Overall Officials: Steven Reynolds, Principal Investigator — Fraser Health Authority
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No